CLINICAL TRIAL: NCT05318131
Title: Sleep, Exercise, Nutrition and Survivorship in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York State Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-00078
Record Dates: First submitted 2022-03-23; First posted 2022-04-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sleep; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Prospective Study (Experimental)
  Interventions: Other: Sleep and Lifestyle Advice Website; Other: Surveys and Sleep Monitors

INTERVENTIONS:
Other: Sleep and Lifestyle Advice Website — Participants will be asked to view a website at least once a week for 3 months (remotely). The website includes information about exercise, nutrition and sleep. Participants will also have a check-in call with a health coach at 6 weeks, and will be sent email newsletters at approximately 1 and 2 months with additional information about sleep, nutrition, and exercise.
Other: Surveys and Sleep Monitors — At baseline and at 3 months, participants will be asked to complete online surveys and to wear an ActiGraph sleep monitor for one week. ActiGraph sleep monitors are wristbands that measure continuous sleep/wake activity information. The recorded ActiGraph data is deidentified and no individual personally identifiable information is collected. A unique serial number identifies each wrist monitor. At the end of the study, participants will also have a telephone exit interview with the study team to provide feedback on their progress during the study and about the website.

SUMMARY:
The primary objectives of this study are to examine sleep, exercise, and nutrition in prostate cancer.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether exposure to a website with recommendations about sleep and lifestyle for patients with prostate cancer and caregivers leads to an improvement in sleep and healthy lifestyle.

ELIGIBILITY:
Inclusion Criteria:

1. Adult U.S. male age >18 with prostate cancer OR
2. Adult U.S. male or female >18 who is a family member/partner/caregiver of a prostate cancer patient AND
3. Telephone and internet access AND
4. Able to read, comprehend, and sign informed consent in English AND
5. Perceived deficits in sleep, nutrition, and/or physical activity

Exclusion Criteria:

1. Age <18 years
2. Not English proficient
3. No or irregular access to the same telephone number and/or mailing address
4. No or less than weekly access to the internet
5. Patients who do not have a diagnosis of prostate cancer
6. Caregivers/family members for a condition other than prostate cancer
7. Mental or cognitive impairment that interferes with ability to provide informed consent
8. Surgery within the past 6 weeks or planned within the next 3 months (must wait until cleared to participate)
9. Other restrictions or upcoming events that affect sleep, physical activity or nutrition (e.g. doctor's orders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Efficiency | Baseline, 3 months
  The study team will use ActiGraph software to calculate device-based measures of sleep efficiency. Sleep efficiency is the ratio of total sleep time (total time spent asleep) to time in bed and is reported as a percentage (total sleep time / time in bed x 100).
Change in Number of Awakenings After Sleep Onset | Baseline, 3 months
  The study team will use ActiGraph software to calculate device-based measure number of awakenings (when a participant wakes up) after sleep onset (the transition from wakefulness into sleep).
Change in Sleep Duration | Baseline, 3 months
  The study team will use ActiGraph software to calculate device-based measures of sleep duration
Change in Sleep Hygiene Index (SHI) Score | Baseline, 3 months
  SHI is a 13-item self-report measure designed to assess the practice of sleep hygiene behaviors. Each item is rated on a five-point scale ranging from 0 (never) to 4 (always). Total scores range from 0 to 52, with a higher score representing poorer sleep hygiene.
Change in Pittsburgh Sleep Quality Index (PSQI) Score | Baseline, 3 months
  PSQI contains 19 self-reported questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points. In all cases, a score "0" indicates no difficulty, while "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points; the higher the score, the more severe the difficulties in all areas.
Change in Insomnia Severity Index Score | Baseline, 3 months
  The Insomnia Severity Index has 7 questions, each rated on a 5-point Likert scale (0-4). The total score range is 0-28; the higher the score, the more severe the insomnia. 0-7 = no clinical significant insomnia, 8-14 = subthreshold insomnia, 15-21 = clinical insomnia (moderate severity), and 22-28 = clinical insomnia (severe)

SECONDARY OUTCOMES:
Change in device-based moderate-vigorous intensity physical activity (MVPA) minutes per day | Baseline, 3 months
  The study team will use ActiGraph's GT3X tri-axial accelerometer and ActiLife software to calculate device-based measures of physical activity. Daily MVPA will be based on least 4 days of at least 10 hours of device wear time. A higher number of minutes of MVPA indicates more physical activity. Among U.S. adults aged 60 years or older, mean number of minutes per day of MVPA ranges from 10.8 to 106.8.
Change in device-based step counts per day | Baseline, 3 months
  The study team will use ActiLife software to calculate step counts per day. Daily steps will be based on at least 4 days of at least 10 hours of device wear time. A higher step count indicates more physical activity. Based on U.S. population samples, normative daily step count ranges are 41 to 12,780 steps for men aged 60 years or older and 55 to 9,735 for women aged 60 years or older.
Change in self-reported total physical activity MET-minutes per day | Baseline, 3 months
  The study team will use the International Physical Activity Questionnaire short form (IPAQ-SF). It will be used to assess time spent in 3 specific types of activity over the previous 7 days: vigorous-intensity activities, moderate-intensity activities, and walking. Time spent in these 3 activity types will be combined to calculate total physical activity minutes per day, a continuous variable with a plausible range of 0 to 960. Then, the study team will apply metabolic equivalents by intensity to calculate total physical activity MET-minutes per day.
Change in Dietary Consumption | Baseline, 3 months
  The study team will use a food frequency questionnaire to measure servings per week of foods. Each food category is measured in never (lowest), once per month, 2-3 times last month, 1 time per week, 2 times per week, 3-4 times per week, 5-6 per week, 1 time per day, 2-3 times per day, 4-5 times per day, and 6+ times per day (highest).

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Loeb, MD MSc, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request for the purposes of an IRB approved scientific research project. Requests should be directed to stacy.loeb@nyulangone.org. To gain access, data requestors will need an IRB approved protocol and to sign a data access agreement.

REFERENCES:
- [Result] Loeb S, Robbins R, Sanchez-Nolasco T, Byrne N, Ruan A, Rivera A, Gupta N, Kenfield SA, Chan JM, Van Blarigan EL, Carter P, Jean-Louis G, Orstad SL. Sleep and health improvement programme (SHIP) for patients with prostate cancer and caregivers. BJUI Compass. 2024 Aug 31;5(10):976-985. doi: 10.1002/bco2.435. eCollection 2024 Oct. PMID 39416756